CLINICAL TRIAL: NCT02037308
Title: The Effects of Beetroot Bread on Postprandial Blood Pressure According to Glu298Asp Polymorphism in the eNOS Gene
Brief Title: Glu298Asp Polymorphism and Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Julie Lovegrove, Professor, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 10/18G; University of Reading (Other: University of Reading)
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2014-01

CONDITIONS: Hypertension
Keywords: Glu298Asp polymorphism; Blood pressure; Plasma NOx; Beetroot
MeSH Terms: conditions — Hypertension | interventions — Bread

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control white bread (Placebo Comparator)
  Interventions: Dietary Supplement: Bread
- Beetroot bread (Experimental)
  Interventions: Dietary Supplement: Bread

INTERVENTIONS:
Dietary Supplement: Bread

SUMMARY:
The Glu298Asp polymorphism has been linked to increased risk of cardiovascular events, proposed to be due to reduced nitric oxide production by eNOS reported in some but not all studies. We hypothesise that beetroot-enriched bread interacts with the Glu298Asp polymorphism of the eNOS gene to lower blood pressure and increase plasma nitrate/nitrite, particularly in carriers of the T allele, which have been associated with lower eNOS activity and increased risk of hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Male
* A signed consent form
* Age 18-64 years
* Body mass index - 18.5-30 kg/m2
* Non-smoking, healthy individuals
* Normal blood pressure at screening (< 150/90)

Exclusion Criteria:

* Subjects with anaemia
* Sufferers of chronic illnesses
* Individuals with food allergies
* People with diabetes
* People with coeliac disease
* Women
* Vegetarians

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2010-06; Primary Completion 2010-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Postprandial blood pressure | 30 minute intervals for a period of 6 hours

SECONDARY OUTCOMES:
Postprandial plasma NOx | 30 minute intervals for a total period of 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Julie Lovegrove, Phd, Principal Investigator — University of Reading
Locations (1):
- Food and Nutritional Sciences, University of Reading, Reading, Berkshire, United Kingdom

REFERENCES:
- [Background] Hobbs DA, Goulding MG, Nguyen A, Malaver T, Walker CF, George TW, Methven L, Lovegrove JA. Acute ingestion of beetroot bread increases endothelium-independent vasodilation and lowers diastolic blood pressure in healthy men: a randomized controlled trial. J Nutr. 2013 Sep;143(9):1399-405. doi: 10.3945/jn.113.175778. Epub 2013 Jul 24. PMID 23884387
- [Background] Hobbs DA, Kaffa N, George TW, Methven L, Lovegrove JA. Blood pressure-lowering effects of beetroot juice and novel beetroot-enriched bread products in normotensive male subjects. Br J Nutr. 2012 Dec 14;108(11):2066-74. doi: 10.1017/S0007114512000190. Epub 2012 Mar 14. PMID 22414688